CLINICAL TRIAL: NCT03170102
Title: Building Capacity of OT Students to Address Children's Mental Health During Fieldwork
Brief Title: Building Capacity of OT Students to Address Children's Mental Health During Fieldwork (OTFW)
Acronym: OTFW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Susan Bazyk, Professor, Cleveland State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FY2016-227
Record Dates: First submitted 2017-05-19; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Education
Keywords: occupational therapy

STUDY DESIGN:
Intervention Model Description: A The study involved a one-group (n=19) mixed methods design using using pretest-posttest surveys and qualitative analysis of written reflections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Building capacity through education (Other): Building capacity process through education - Occupational therapy students participate in online webinars and discussions following completion of readings.
  Interventions: Other: Building capacity through education

INTERVENTIONS:
Other: Building capacity through education — Participants engaged in 2 webinars and 3 online discussions following reading selected material.

SUMMARY:
The study involved a one-group (n=19) mixed methods design using using pretest-posttest surveys and qualitative analysis of written reflections was used to explore the meaning and outcomes of participation in the building capacity process.

DETAILED DESCRIPTION:
To explore the meaning and outcomes of a four-month building capacity process designed to promote knowledge translation of a public health approach to mental health with children and youth among occupational therapy students completing a Level II Fieldwork experience in school-based practice.The study involved a one-group (n=19) mixed methods design using using pretest-posttest surveys and qualitative analysis of written reflections was used to explore the meaning and outcomes of participation in the building capacity process.The building capacity process expanded student knowledge of a public health approach to mental health resulting in increased awareness and application of embedded strategies addressing mental health during a Level II Fieldwork experience in a school settings.

ELIGIBILITY:
Inclusion Criteria:

* Occupational therapy (OT) students completing a Level II Fieldwork experience during Fall 2016 in a school setting
* OT students meeting the above criteria who agree to participate in the study

Exclusion Criteria:

- OT students completing a FW experience in settings other than schools during Fall 2016

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in knowledge, beliefs, and actions regarding addressing children's mental health in a school-based fieldwork experience | 2 weeks
  20 questions using Likert Scale responses

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bazyk, PhD, Principal Investigator — Cleveland State University

IPD SHARING:
Plan to Share IPD: No